CLINICAL TRIAL: NCT06001307
Title: HIV Risk Reduction Intervention for Transwomen With Intimate Partner Victimization
Brief Title: Supporting Trans Affirmation, Relationships, and Sex, Phase 3
Acronym: STARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); The University of Akron (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2002002648; 1R34MH119968-01A1 (NIH)
Record Dates: First submitted 2023-08-04; First posted 2023-08-21 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: HIV; Violence, Gender-Based; Violence, Domestic; Risk Reduction Behavior
Keywords: LGBTQ; HIV Prevention; Transgender research; Peer counseling; Intimate Partner Violence (IPV); PrEP
MeSH Terms: conditions — Risk Reduction Behavior | interventions — Association; Sex

STUDY DESIGN:
Intervention Model Description: The methodological approach includes a 2-arm trial of Project STARS vs. a time matched, attention-controlled comparison group, with up to n=20 per arm (total Phase 3 sample size = up to 40 participants enrolled and randomized). The study is intended to evaluate the impacts of STARS on the specified outcomes.
Who Masked: Outcomes Assessor
Masking Description: All research staff conducting participant assessments will remain blinded to group assignment. Randomization procedures will be conducted by a high level researcher (co-investigator responsible for clinical supervision).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Program STARS (Supporting Trans Affirmation, relationships, and Sex) (Experimental): STARS is an HIV prevention intervention for trans women/femmes with recent intimate partner violence (IPV). Delivered by peer counselors, STARS consists of two one-hour sessions held one week apart and two brief 20-30 minute booster sessions held two- and four-weeks after the 2nd hour long session. Requirements for peer counselors include identifying as trans women or trans feminine and having leadership roles in the trans community.
  STARS is an empowerment-based intervention that integrates trauma-informed and gender affirmation approaches. The first session emphasizes education and discussion around HIV and IPV, as well as the interaction between IPV and HIV risk. The second session focuses on identifying partners where HIV/IPV risk exists and developing an empowerment plan to address those risks. Participants create an empowerment plan in session 2 and this plan is reviewed and updated in the booster sessions.
  Interventions: Behavioral: Program STARS (Supporting Trans Affirmation, relationships, and Sex)
- Relaxation and Stress Reduction (Active Comparator): The Relaxation and Stress Reduction Program is structured to mirror STARS (time matched, attention-controlled). Delivered by peer counselors, the Relaxation and Stress Reduction Program consists of two one-hour sessions held one week apart and two brief 20-30 minute booster sessions held two- and four-weeks after the 2nd hour long session. Requirements for peer counselors include identifying as trans women or trans feminine and having leadership roles in the trans community.
  The relaxation and stress reduction protocol is an attention and time-matched control condition. The intervention focuses on providing both education and opportunities to practice various relaxation strategies. In addition, education is provided on healthy eating as an additional tool for reducing stress. Booster sessions focus on providing participants with additional practice of relaxation strategies.
  Interventions: Behavioral: Relaxation and Stress Reduction

INTERVENTIONS:
Behavioral: Program STARS (Supporting Trans Affirmation, relationships, and Sex) — See description to the left.
  Arms: Program STARS (Supporting Trans Affirmation, relationships, and Sex)
Behavioral: Relaxation and Stress Reduction — See description to the left.
  Arms: Relaxation and Stress Reduction

SUMMARY:
The purpose of this clinical trial is to evaluate and test a newly developed gender-affirming intervention that addresses the dual and interconnected risks of HIV and intimate partner victimization (IPV) among transgender women (TW). The main questions it aims to answer are: (1) will the study intervention reduce HIV risk within the context of IPV and related risk factors (e.g., substance use and PTSD); (2) will STARS improve primary prevention behaviors, such as condom use, pre-exposure prophylaxis (PrEP) use, and repeat HIV testing; and (3) what are the mechanisms of change relevant to the theoretical foundations of the intervention, including gender affirmation, empowerment, and self-efficacy. The findings from this study will provide the necessary groundwork to examine the efficacy of this combined HIV-IPV intervention in a future, large-scale clinical trial.

There are several components to this research study:

* First, participants will be asked to complete a series of screening interviews/questionnaires to determine eligibility, including completing a HIV test.
* If eligible, participants will then take part in a 2-3 hour baseline assessment consisting of both interviewer administered questionnaires as well as self-administered surveys.
* Participants will then be randomly assigned to one of two treatment conditions: (1) a newly developed gender affirming intervention, known as Program STARS (Supporting Trans Affirmation, relationships, and Sex) or (2) a time-matched, attention-controlled program that offers free training in relaxation and stress reduction techniques (a.k.a., the comparison group). Both interventions offer unique components and the researchers do not yet know the impact the programs may have on participants' overall well-being.
* Participants randomized to Project STARS, will be invited to complete a semi-structured exit interview (lasting 60-90 min.) after the completion of the program.
* This clinical trial has three follow-up assessments: (1) post-intervention (i.e., after the peer-counseling programs are complete); (2) at 4-months follow-up; and (3) at 6-months follow-up. The follow-up assessments are structured the same way as the baseline assessment and are estimated to take around 1-2 hours.

The total study involvement for this clinical trial is estimated to take approximately 10 to 12 hours over the course of six months.

DETAILED DESCRIPTION:
Transgender women (TW) are among the populations most heavily affected by HIV in the United States (US), with nearly 1 in 5 TW living with HIV. The risk for HIV in TW often occurs in the context of intimate partner relationships. Moreover, in the context of these partnerships, TW are at elevated risk for intimate partner victimization (IPV). There is a strong link between IPV and HIV risk. IPV risk is amplified in TW who have a history of IPV or are in an abusive primary relationship. Thus, IPV and HIV as well as other sexually transmitted infections (STIs) are interconnected public health problems facing TW. Despite the dual and interconnected risks of HIV and IPV among TW, there are few empirically based HIV prevention interventions that target TW and none that target HIV risks related to IPV in this population.

This overall research study is a 3-phase project (NIH R34MH119968). In Phase 1, researchers conducted focus groups with TW and community-based service providers to identify specific strategies for a brief health educational counseling intervention to support safety and HIV risk reduction among TW who have experienced recent IPV and HIV risk. Phase 1 data collection activities and preliminary analyses have been completed, and a full draft intervention protocol was produced based on Phase 1 findings.

Phase 2 of this study involved conducting an open pilot trail (OP) of the full draft intervention protocol with 5 participants, using quantitative (i.e. surveys) and qualitative (i.e. individual interviews) methods to gain experience delivering the protocol and obtaining critical feedback on the intervention protocol, procedures and assessments. This knowledge has informed finalizing the intervention and assessment protocols, which will be used in the subsequent and final Phase 3 of the study.

Phase 3 (the clinical trial registered here), involves conducting a pilot, two-arm Randomized Control Trial (RCT) to evaluate the program's ability to increase knowledge of HIV and HIV risk factors and reduce risk of intimate partner victimization among participants. The two treatment conditions used in this clinical trial are: (1) a newly developed gender affirming intervention, known as Program STARS (Supporting Trans Affirmation, relationships, and Sex) - detailed below and (2) a time-matched, attention-controlled program that offers free training in relaxation and stress reduction techniques (a.k.a., the comparison group).

Participants will first complete a multi-step screening process to determine eligibility. If eligible, enrolled participants will then complete a 2-3 hour baseline assessment that can be conducted in-person or over Zoom. Assessments consist of interviewer administered safety measures as well as self-report online questionnaires. After completing the baseline assessment, participants will be randomly assigned to one of the two intervention arms. Assessments will also be conducted post-intervention as well as at 4-months and 6-months follow up. Participants who were randomized to the study intervention arm (i.e., the STARS Program) will also be invited to complete a 60-90 minute semi-structured exit interview via Zoom to provide qualitative feedback on the program.

The overall purpose of this study is to develop a brief intervention that concurrently targets HIV and IPV risk, as well as addresses inter-related risks of HIV and IPV (e.g., substance use and PTSD) for TW - referred to as Supporting Transwomen Affirmation, Relationships and Sex (STARS). Program STARS will:

* Be based on the Gender Affirmation Framework, which emphasizes interpersonal processes to positively affirm the identities and unique needs of TW.
* Integrate a trauma-informed empowerment approach.
* Include gender-affirming and empowering HIV prevention counseling that addresses HIV risk within the context of IPV and related risk factors (e.g., substance use and PTSD), and a range of HIV risk reduction options.
* Provide TW with behavioral skills and resources for addressing IPV and maximizing personal safety.

The aims of this treatment development research are to:

1. Develop a behavioral intervention manual that addresses the specific and unique HIV prevention needs of TW with IPV, and that uses a gender-affirmative, empowering, and trauma-informed approach; and
2. Evaluate the feasibility, acceptability, safety, and initial effects of STARS through three phases of intervention development.

Researchers are primarily interested in exploring the pattern of results for any evidence of support for the intervention's influence on the primary and secondary outcomes, which are listed below.

Primary Outcomes:

1. Composite Risk for HIV (CR-HIV) is a binary indicator of any HIV risk (e.g., yes=1 vs. no=0), which is an algorithm based on whether the participant:

   * report condomless anal sex with a HIV serodiscordant or status-unknown primary or other partner in the past 3 months;
   * is using PrEP;
   * is in a monogamous partnership with an HIV-uninfected partner or an ;
   * is in a monogamous partnership with an HIV-infected partner who is virally suppressed.
   * If participants are not certain about the latter two indicators, they are coded as having HIV risk according to this algorithm.
2. IPV frequency will be assessed with:

   * The Composite Abuse Scale revised short form (CASr-SF).and
   * A trans-specific IPV Scale (T-IPV Scale; Peitzmeier et al, in press) that assesses IPV unique to TW (e.g., being forced not pursuing aspects of gender transition that you wanted).
3. IPV safety will be assessed with the:

   * Measure Of Victim Empowerment Related to Safety (MOVERS; Goodman et al., 2015), which is a 13-item scale that measures IPV survivors' safety-related psychosocial skills and efficacy and expectations of support, as well as the extent to which survivors feel that their efforts to achieve safety might create new difficulties.

Secondary Outcomes:

* Biologically determined STI diagnoses, including HIV - The research staff will work with participants to find gender-affirming health care clinics in their area that provide free or low-cost STI and HIV testing. Participants will be encouraged to get tested for STIs as part of the research study; however, STI testing is not a requirement for participation. HIV self-test kits will be mailed to willing participants and the research staff will walk participants through testing procedures as well as post-test result counseling (as needed) over Zoom or in-person.
* Self-reported discrete behavioral risk indicators: CAS, multiple and concurrent partnerships, partners' HIV status, monogamy and sexual agreements, substance use including injection drug use, HIV testing behaviors (including self-testing) and knowledge, intentions to use PrEP, PrEP uptake, use of any HIV prevention services, and use of any additional IPV-related services/resources.

Long-term aim: The findings from this R34 intervention development study will provide the groundwork to examine the efficacy of STARS in a future, large-scale clinical trial, which can be readily implemented in real-world settings.

Dissemination

* Throughout the study, researchers will disseminate process reports and descriptive summaries of the findings to colleagues at social service and medical/health agencies with whom we established MOUs.
* As data are evaluated, researchers will prepare brief reports describing the major findings from the study which we will share with our community partners, HIV prevention and IPV scientists, and TW health and advocacy organizations through publications and presentations at professional conferences.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old;
* Assigned male at birth but identify as female, transgender, or transfeminine;
* Endorse at least one IPV incident during the previous 12 months based on the trans-specific IPV Scale (T-IPV Scale; Peitzmeier et al, in press);
* Report at least one instance of condomless anal sex in the last 6 months.

Exclusion Criteria:

* Have been diagnosed with HIV or test positive for HIV.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Assigned male at birth and identify as female, transgender, or transfeminine
Enrollment: 37 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shufang Sun, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Following data collection, cleaning, and analysis, we plan to publish deidentified quantitative data at an open science data repository (e.g., Open Science Framework). De-identified qualitative data will be available upon request to the study PI.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available sometime in during Summer 2024 and will be available for the duration of staff funding.

REFERENCES:
- [Derived] Guy AA, Chen CA, McCarthy-Belash N, Kang TK, Kolbasov LA, Gregory R, Scott T, Garcia J, Banson J, Zlotnick C, Operario D, Johnson DM, Sun S. Mixed methods trial of a peer intervention for HIV and partner victimization in transgender women. J Couns Psychol. 2025 Nov 6:10.1037/cou0000832. doi: 10.1037/cou0000832. Online ahead of print. PMID 41196739

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Program STARS (Supporting Trans Affirmation, relationships, and Sex) | Relaxation and Stress Reduction
Started | 19 | 18
Post-intervention Assessment | 19 | 17 (In the control arm, 1 participant was lost to follow-up.)
4-month Follow-up Assessment (In the STARS arm, 1 participant was lost to follow-up; and 1 participant missed the assessment window. In the control arm, 2 participants were lost to follow-up; and 5 participants missed their assessment window. Participants who missed their 4-month follow-up assessment windows were still invited to complete the 6-month follow-up assessments.) | 17 | 11
6-month Follow-up Assessment (In the STARS arm, 1 participant was lost to follow-up. In the control arm, 2 participants was lost to follow-up.) | 18 | 16
Completed | 18 | 16
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Program STARS (Supporting Trans Affirmation, Relationships, and Sex) | Relaxation and Stress Reduction | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.42 (8.88) | 35.28 (9.20) | 33.81 (9.02)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Feminine/femme or transfeminine | 4 | 6 | 10
  Māhū, or muxe, or two spirit | 2 | 0 | 2
  Non-binary | 1 | 1 | 2
  Woman or Transgender Woman | 10 | 11 | 21
  None of these describe me | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Multiracial participants were able to select multiple race/ethnicity
  Participants
    American Indian or Alaska Native | 2 | 1 | 3
    Asian American and Pacific Islander | 0 | 3 | 3
    Black/African American | 2 | 0 | 2
    White/Caucasian | 16 | 16 | 32
    Other | 3 | 0 | 3
    Hispanic or Latina | 3 | 4 | 7
Frequency of past-year IPV [Mean (Standard Deviation); unit: Events] | 14.32 (11.09) | 9.67 (10.26) | 12.06 (10.81)
PTSD symptoms [Mean (Standard Deviation); unit: Scores on a scale] — PTSD symptoms were evaluated using the PTSD Checklist for DSM-5, a 20-item measure that assesses symptom frequency in the past month on a five-point Likert scale (0 = "Not at all" to 4 = "Extremely"). The total score is calculated by summing the responses for all 20 items, resulting in a score between 0 and 80. A higher total score indicates more severe PTSD symptoms.
  Scores on a scale | 41.32 (12.29) | 33.94 (13.87) | 37.73 (13.43)
Depressive Symptoms [Mean (Standard Deviation); unit: Scores on a scale] — Depressive symptoms were evaluated using the Center of Epidemiologic Studies Depression Scale-10 (CESD-10). The measure consists of 10 items that asked about feelings or behaviors related to depressive symptoms on a four-point Likert scale (0-3). Items 5 and 8 were first reverse coded, and all points were summed to create a total score ranging from 0 to 30, with higher scores representing greater degrees of depressed mood.
  Scores on a scale | 15.53 (4.83) | 12.90 (5.79) | 14.26 (5.41)
Total number of receptive condomless anal sex acts with any HIV transmission risk [Mean (Standard Deviation); unit: Events] — The total number of receptive condomless anal sex acts with any HIV transmission risk was calculated by summing the number of receptive anal sex acts in which no prevention method (i.e., condom, PrEP) was used over the last 60 days.
  Events | 0.16 (0.69) | 0.83 (2.36) | 0.49 (1.73)
Composite Risk for HIV (CR-HIV) [Count of Participants; unit: Participants] — Composite Risk for HIV calculates a binary indicator (0=No, 1=Yes) of risk for HIV acquisition based on the following questions:
  1. Do they report condomless anal sex with a HIV serodiscordant or status-unknown primary or other partner in the past 6 months? (If yes, move on to question #2; If no, 0)
  2. Is the participant using PrEP? (If yes, 0; If no, move onto question #3)
  3. Is the participant in a monogamous partnership with an HIV-uninfected partner or an HIV-infected partner who is virally suppressed? (If yes, 0; If no, 1) Number of participants at risk is reported for each arm.
  Participants | 1 | 3 | 4
Intimate Partner Violence (IPV) Frequency [Mean (Standard Deviation); unit: Scores on a scale] — Intimate Partner Violence (IPV) Frequency was measured using the Composite Abuse Scale Revised-Short Form (CASr-SF), a 15-item scale. For each item, participants answer if the type of abuse occurred and how often from, "Not in the past 2 months (0)" to "Daily/ almost daily (5)." Total score was calculated by summing all items, which could range from 0 to 75 with higher scores indicate higher frequency and severity of IPV.
  Scores on a scale | 4.16 (4.73) | 3.06 (4.21) | 3.63 (4.46)
Intimate Partner Violence Frequency: Transgender-specific IPV scale (T-IPV) [Mean (Standard Deviation); unit: Scores on a scale] — IPV frequency is assessed using the trans-specific IPV scale (T-IPV), a 4-item scale that screens for IPV among transgender individuals. Participants reponsded to statements covering the presence of controlling behaviors and psychological abuse tactics (No=0; Yes=1). Scores range from 0 to 4, with higher scores indicating higher frequency of recent T-IPV.
  Scores on a scale
    Past year | 1.16 (1.74) | 0.67 (1.14) | 0.92 (1.48)
    Past two months | 0.16 (0.50) | 0.28 (0.83) | 0.22 (0.67)
Intimate Partner Violence Safety: Measure Of Victim Empowerment Related to Safety (MOVERS) [Mean (Standard Deviation); unit: Scores on a scale] — MOVERS is a 13-item scale designed to assess empowerment related to safety among IPV survivors. Participants rate each item on a five-point Likert scale (1 = Never true to 5 = Always true). For each participant, the mean score across all 13 items was calculated (score range: 1-5). The scale includes 3 subscales: Internal Tools, Expectations of Support, and Trade-Offs. Scores for each subscale were computed as the mean score of the items corresponding to that subscale (score range: 1-5 for all subscales). For both the composite scale and subscales, higher scores indicate greater empowerment.
  Scores on a scale
    Composite score | 3.55 (0.48) | 3.59 (0.60) | 3.57 (0.54)
    Internal Tools subscale | 3.47 (0.68) | 3.53 (0.60) | 3.50 (0.63)
    Expectations of Support subscale | 3.28 (0.75) | 3.38 (0.92) | 3.33 (0.83)
    Trade-Offs subscale | 3.91 (0.70) | 3.87 (0.67) | 3.89 (0.68)

OUTCOME MEASURES:

1. Primary Outcome: Composite Risk for HIV (CR-HIV)
Description: Composite Risk for HIV (CR-HIV) calculates a binary indicator (0=No, 1=Yes) of a participant's risk for HIV acquisition using an algorithm based on the following questions:
  1. Do they report condomless anal sex with a HIV serodiscordant or status-unknown primary or other partner in the past 6 months? (If yes, move on to question #2; If no, 0)
  2. Is the participant using PrEP? (If yes, 0; If no, move onto question #3)
  3. Is the participant in a monogamous partnership with an HIV-uninfected partner or an HIV-infected partner who is virally suppressed? (If yes, 0; If no, 1) *If participants are not certain about their partner's HIV status or viral suppression status in the last question, they are coded as having HIV risk according to this algorithm.
  The total number of participants at risk for HIV acquisition for each arm is reported.
Time Frame: Post-intervention, 4-month follow-up, and 6-month follow-up
Population: 3 participants were lost to attrition. In the STARS arm, 1 participant was lost after the post-intervention assessment. In the control arm, 1 participant was lost after the baseline assessment, and 1 participant was lost after the post-intervention assessment.
  At 4-month follow-up, 1 participant in the STARS arm and 5 in the control arm missed the assessment window. However, these participants still completed the 6-month follow-up assessment and were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Program STARS (Supporting Trans Affirmation, relationships, and Sex) | Relaxation and Stress Reduction
Number analyzed (Participants) | 19 | 18
Participants
  Post-intervention: number analyzed (Participants) | 19 | 17
  Post-intervention | 0 | 1
  4-month follow-up: number analyzed (Participants) | 17 | 11
  4-month follow-up | 9 | 1
  6-month follow-up: number analyzed (Participants) | 18 | 16
  6-month follow-up | 0 | 1

2. Primary Outcome: Intimate Partner Violence (IPV) Frequency: Composite Abuse Scale Revised Short Form (CASr-SF)
Description: Intimate Partner Violence (IPV) Frequency was measured using the Composite Abuse Scale Revised-Short Form (CASr-SF), a 15-item scale. For each item, participants answer if the type of abuse occurred and how often from, "Not in the past 2 months (0)" to "Daily/ almost daily (5)." Total score was calculated by summing all items, which could range from 0 to 75 with higher scores indicate higher frequency and severity of IPV.
Time Frame: Post-intervention, 4-month follow-up, and 6-month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Program STARS (Supporting Trans Affirmation, relationships, and Sex) | Relaxation and Stress Reduction
Number analyzed (Participants) | 19 | 18
Scores on a scale
  Post-intervention: number analyzed (Participants) | 19 | 17
  Post-intervention | 2.37 (4.27) | 1.18 (2.38)
  4-month follow-up: number analyzed (Participants) | 17 | 11
  4-month follow-up | 1.06 (2.93) | 0.82 (2.09)
  6-month follow-up: number analyzed (Participants) | 18 | 16
  6-month follow-up | 0.22 (0.65) | 0.63 (1.62)

3. Primary Outcome: Intimate Partner Violence (IPV) Frequency: Transgender-Specific Intimate Partner Violence (T-IPV) Scale
Description: IPV frequency is assessed using the trans-specific IPV scale (T-IPV), a 4-item scale that screens for IPV among transgender individuals. Participants reponsded to statements covering the presence of controlling behaviors and psychological abuse tactics (No=0; Yes=1). Scores range from 0 to 4, with higher scores indicating higher frequency of recent T-IPV.
Time Frame: Post-intervention, 4-month follow-up, and 6-month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Program STARS (Supporting Trans Affirmation, relationships, and Sex) | Relaxation and Stress Reduction
Number analyzed (Participants) | 19 | 18
Scores on a scale
  Post-intervention: number analyzed (Participants) | 19 | 17
  Post-intervention | 0 (0) | 0 (0)
  4-month follow-up: number analyzed (Participants) | 17 | 11
  4-month follow-up | 0 (0) | 0 (0)
  6-month follow-up: number analyzed (Participants) | 18 | 16
  6-month follow-up | 0 (0) | 0.06 (0.25)

4. Primary Outcome: Intimate Partner Violence (IPV) Safety: Measure Of Victim Empowerment Related to Safety (MOVERS)
Description: MOVERS is a 13-item scale designed to assess empowerment related to safety among IPV survivors. Participants rate each item on a five-point Likert scale (1 = Never true to 5 = Always true). For each participant, the mean score across all 13 items was calculated (score range: 1-5). The scale includes 3 subscales: Internal Tools, Expectations of Support, and Trade-Offs. Scores for each subscale were computed as the mean score of the items corresponding to that subscale (score range: 1-5 for all subscales). For both the composite scale and subscales, higher scores indicate greater empowerment.
Time Frame: Post-intervention, 4-month follow-up, and 6-month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Program STARS (Supporting Trans Affirmation, relationships, and Sex) | Relaxation and Stress Reduction
Number analyzed (Participants) | 19 | 18
Scores on scale
  Post-intervention (Composite): number analyzed (Participants) | 19 | 17
  Post-intervention (Composite) | 3.65 (0.63) | 3.46 (0.74)
  4-month follow-up (Composite): number analyzed (Participants) | 17 | 11
  4-month follow-up (Composite) | 3.82 (0.51) | 3.61 (0.51)
  6-month follow-up (Composite): number analyzed (Participants) | 18 | 16
  6-month follow-up (Composite) | 3.77 (.57) | 3.73 (.49)
  Post-intervention (Internal Tools subscale): number analyzed (Participants) | 19 | 17
  Post-intervention (Internal Tools subscale) | 3.69 (0.74) | 3.43 (0.85)
  4-month follow-up (Internal Tools subscale): number analyzed (Participants) | 17 | 11
  4-month follow-up (Internal Tools subscale) | 3.94 (0.69) | 3.76 (0.70)
  6-month follow-up (Internal Tools subscale): number analyzed (Participants) | 18 | 16
  6-month follow-up (Internal Tools subscale) | 3.95 (0.52) | 3.65 (0.75)
  Post-intervention (Expectations of Support subscale): number analyzed (Participants) | 19 | 17
  Post-intervention (Expectations of Support subscale) | 3.45 (1.03) | 3.35 (1.03)
  4-month follow-up (Expectations of Support subscale): number analyzed (Participants) | 17 | 11
  4-month follow-up (Expectations of Support subscale) | 3.63 (0.82) | 3.57 (0.66)
  6-month follow-up (Expectations of Support subscale): number analyzed (Participants) | 18 | 16
  6-month follow-up (Expectations of Support subscale) | 3.51 (0.95) | 3.66 (0.83)
  Post-intervention (Trade-Offs subscale): number analyzed (Participants) | 19 | 17
  Post-intervention (Trade-Offs subscale) | 3.81 (0.75) | 3.61 (0.76)
  4-month follow-up (Trade-Offs subscale): number analyzed (Participants) | 17 | 11
  4-month follow-up (Trade-Offs subscale) | 3.88 (0.95) | 3.52 (0.90)
  6-month follow-up (Trade-Offs subscale): number analyzed (Participants) | 18 | 16
  6-month follow-up (Trade-Offs subscale) | 3.85 (0.91) | 3.88 (0.75)

5. Primary Outcome: Feasibility of Online STARS as Measured by Recruitment Rates
Description: One measure of feasibility will be participant recruitment rates.
Time Frame: During recruitment period of study, up to 4 months
Population: Overall Number of Participants Analyzed represents number of participants screened for study interest prior to enrollment.
Measure: Count of Participants; unit: Participants
Groups:
- Pre-randomization: First, the recruitment rate was calculated by comparing the total number of participants screened eligible to those who were successfully enrolled in the study.
Arm/Group | Pre-randomization
Number analyzed (Participants) | 98
Participants | 37

6. Primary Outcome: Feasibility of Online STARS as Measured by Retention Rates.
Description: One measure of feasibility will be participant retention rates, as measured by engagement/completion of the interventions.
Time Frame: Post-intervention, 4-month follow-up, and 6-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Program STARS (Supporting Trans Affirmation, relationships, and Sex) | Relaxation and Stress Reduction
Number analyzed (Participants) | 19 | 18
Participants
  Post-intervention | 19 | 17
  4-month follow-up | 17 | 11
  6-month follow-up | 18 | 16

7. Primary Outcome: Acceptability of Online STARS as Measured by the Client Satisfaction Questionnaire
Description: One measure of acceptability will be via acceptability ratings using the validated 8-item Client Satisfaction Questionnaire (CSQ-8). Participants rated each item on a four-point Likert scale. For each participant, the mean score across all 8 items was calculated (score range: 1-4), with higher values indicating higher satisfaction.
Time Frame: Post-intervention
Population: In the control arm, 1 participant was lost to follow-up after the baseline assessment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Program STARS (Supporting Trans Affirmation, relationships, and Sex) | Relaxation and Stress Reduction
Number analyzed (Participants) | 19 | 17
Scores on a scale | 3.29 (.48) | 2.95 (.8)

8. Other Pre Specified Outcome: Participants Reporting Instances of IPV
Time Frame: Post-intervention, 4-month follow-up, 6-month follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Program STARS (Supporting Trans Affirmation, relationships, and Sex) | Relaxation and Stress Reduction
Number analyzed (Participants) | 19 | 18
Participants
  Post-intervention: number analyzed (Participants) | 19 | 17
  Post-intervention | 7 | 5
  4-month follow-up: number analyzed (Participants) | 17 | 11
  4-month follow-up | 5 | 3
  6-month follow-up: number analyzed (Participants) | 18 | 16
  6-month follow-up | 2 | 3

9. Other Pre Specified Outcome: Depressive Symptoms
Description: Depressive symptoms were evaluated using the Center of Epidemiologic Studies Depression Scale-10 (CESD-10). The measure consists of 10 items that asked about feelings or behaviors related to depressive symptoms on a four-point Likert scale (0-3). Items 5 and 8 were first reverse coded, and all points were summed to create a total score ranging from 0 to 30, with higher scores representing greater degrees of depressed mood.
Time Frame: Post-intervention, 4-month follow-up, 6-month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Program STARS (Supporting Trans Affirmation, relationships, and Sex) | Relaxation and Stress Reduction
Number analyzed (Participants) | 19 | 18
Scores on a scale
  Post-intervention | 13.63 (6.32) | 12.47 (5.54)
  4-month follow-up: number analyzed (Participants) | 17 | 11
  4-month follow-up | 12.29 (5.60) | 13.27 (6.17)
  6-month follow-up: number analyzed (Participants) | 18 | 16
  6-month follow-up | 13.11 (5.88) | 13.19 (7.58)

10. Other Pre Specified Outcome: PTSD Symptoms: PTSD Checklist for DSM-5 (PCL-5)
Description: PTSD symptoms were evaluated using the PTSD Checklist for DSM-5, a 20-item measure that assesses symptom frequency in the past month on a five-point Likert scale (0 = "Not at all" to 4 = "Extremely"). The total score is calculated by summing the responses for all 20 items, resulting in a score between 0 and 80. A higher total score indicates more severe PTSD symptoms.
Time Frame: Post-intervention, 4-month follow-up, and 6-month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Program STARS (Supporting Trans Affirmation, relationships, and Sex) | Relaxation and Stress Reduction
Number analyzed (Participants) | 19 | 18
Scores on a scale
  Post-intervention: number analyzed (Participants) | 19 | 17
  Post-intervention | 32.68 (16.13) | 26.59 (10.74)
  4-month follow-up: number analyzed (Participants) | 17 | 11
  4-month follow-up | 30.76 (16.04) | 27.91 (16.91)
  6-month follow-up: number analyzed (Participants) | 18 | 16
  6-month follow-up | 26.83 (14.86) | 31.31 (19.57)

11. Secondary Outcome: Total Number of Receptive Condomless Anal Sex Acts With Any HIV Transmission Risk
Description: The total number of receptive condomless anal sex acts with any HIV transmission risk was calculated by summing the number of receptive anal sex acts in which no prevention method (i.e., condom, PrEP) was used over the last 60 days.
Time Frame: Post-intervention, 4-months follow-up, 6-months follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Program STARS (Supporting Trans Affirmation, relationships, and Sex) | Relaxation and Stress Reduction
Number analyzed (Participants) | 19 | 18
Events
  Post-intervention: number analyzed (Participants) | 19 | 17
  Post-intervention | 0 (0) | 0.5 (.24)
  4-month follow-up: number analyzed (Participants) | 17 | 11
  4-month follow-up | 0 (0) | 1.45 (4.82)
  6-month follow-up: number analyzed (Participants) | 18 | 16
  6-month follow-up | 0 (0) | .25 (1)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 6 months
Arm/Group | Program STARS (Supporting Trans Affirmation, relationships, and Sex) | Relaxation and Stress Reduction
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 5/19 | 0/18
Other Adverse Events (participants affected / at risk) | 1/19 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Program STARS (Supporting Trans Affirmation, relationships, and Sex) (N=19) | Relaxation and Stress Reduction (N=18)
Serious/life threatening IPV (Social circumstances) | 3 | NA
Rape or attempted rape (Social circumstances) | 4 | NA — Indicated by item 8 on CAS-SF
Hospitalization (Psychiatric disorders) | 1 | NA — Mental Health
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Program STARS (Supporting Trans Affirmation, relationships, and Sex) (N=19) | Relaxation and Stress Reduction (N=18)
Sexual assault other than rape or attempted rape (Social circumstances) | 1 | NA — Indicated by items 3, 6, 7 on CAS-SF or any increase in DA-5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT06001307/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT06001307/SAP_001.pdf
  • Informed Consent Form (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT06001307/ICF_002.pdf